CLINICAL TRIAL: NCT07180953
Title: Route of Dexamethasone Administration in iPACK and ACB for Total Knee Replacement: A Randomized Trial
Brief Title: Impact of Dexamethasone Route on Pain and Inflammation in iPACK With ACB for Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02/20025
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee; Knee Pain Chronic; Arthropathy of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Placebo Comparator): iPACK block with ACB
  Interventions: Drug: NaCl 0.9%
- iv DEX (Active Comparator): iPACK block with ACB + iv Dexamethasone
  Interventions: Drug: Dexamethasone 4mg
- pn DEX (Active Comparator): iPACK block with ACB + perineural Dexamethasone
  Interventions: Drug: Dexamethasone 4mg

INTERVENTIONS:
Drug: NaCl 0.9% — iPACK block with Adductor Canal Block (2 x 20ml 0.2% ropivacaine + 1ml 0.9% NaCl) + 2ml 0.9% NaCl iv
  Arms: Control
Drug: Dexamethasone 4mg — iPACK block with Adductor Canal Block (2 x 20ml 0.2% ropivacaine + 1ml 0.9% NaCl) + 4mg Dexamethasone iv
  Other Names: iv Dexamethasone
  Arms: iv DEX
Drug: Dexamethasone 4mg — iPACK block with Adductor Canal Block (2 x 20ml 0.2% ropivacaine + 2mg Dexamethasone) + 2ml 0.9% NaCl iv
  Arms: pn DEX

SUMMARY:
"The Effect of Dexamethasone Administration Route on Pain and Inflammatory Response in iPACK With ACB for Total Knee Arthroplasty" - written in plain language according to ClinicalTrials.gov standards:

The goal of this clinical trial is to learn how the route of dexamethasone administration (either through the vein or nerve block) affects pain and inflammation in people having total knee replacement surgery. All participants will receive two types of nerve blocks before surgery: an iPACK block and an adductor canal block (ACB), which help control pain after the operation.

The main questions the study aims to answer are:

Does injecting dexamethasone into the nerve block reduce pain more effectively than giving it by vein? Which method leads to a lower inflammatory response after surgery? Researchers will compare the two groups to see which route offers better pain relief and less swelling after knee surgery.

Participants will:

Be randomly assigned to receive dexamethasone either in the nerve block or by IV Receive standard care for total knee replacement Rate their pain and have blood tests after surgery to measure inflammation

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for total knee arthroplasty
* patients aged >65 and <100 years
* patients can provide informed consent
* patients can reliably report symptoms to the research team

Exclusion Criteria:

* inability to provide first-party consent due to cognitive impairment or a
* language barrier
* infection at the site of the regional block,
* coagulation disorders,
* immunodeficiency,
* American Society of Anesthesiologists (ASA) physical status of IV or higher,
* history of regular steroid medication.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | Time Frame: 48 hours after surgery
  Time to first rescue analgesia

SECONDARY OUTCOMES:
Total opioid consumption | 48 hours after surgery
  Total opioid consumption (mg) converted to morphine milligram equivalents (MME)
NRS | 4 hours after surgery
  umeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 8 hours after surgery
  umeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 12 hours after surgery
  umeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 24 hours after surgery
  umeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NRS | 48 hours after surgery
  umeric Rating Scale (NRS), ranging from 0 ("no pain") to 10 ("the worst pain imaginable")
NLR | 12 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 24 hours after surgery
  Neutrophil-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 12 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 24 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 4 hours after surgery
  Quadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale, where higher scores indicate better muscle strength
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 8 hours after surgery
  Quadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale, where higher scores indicate better muscle strength
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 12 hours after surgery
  Quadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale, where higher scores indicate better muscle strength
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 24 hours after surgery
  Quadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale, where higher scores indicate better muscle strength
Quadriceps muscle strength assessed using medical research council scale [range 0:5] | 48 hours after surgery
  Quadriceps muscle strength, including knee extension and hip adduction, will be evaluated using the Medical Research Council (MRC) muscle strength grading scale, where higher scores indicate better muscle strength
Nerve damage | 12 hours after surgery
  Nerve damage assessment will be performed using the following grading scale:
  N0 - No nerve damage N1 - Minor: sensory paresthesia N2 - Major: complete sensory anesthesia N3 - Complete: complete motor deficit with or without paresthesia N4 - CRPS: Complex Regional Pain Syndrome
Nerve damage | 24 hours after surgery
  Nerve damage assessment will be performed using the following grading scale:
  N0 - No nerve damage N1 - Minor: sensory paresthesia N2 - Major: complete sensory anesthesia N3 - Complete: complete motor deficit with or without paresthesia N4 - CRPS: Complex Regional Pain Syndrome
Nerve damage | 48 hours after surgery
  Nerve damage assessment will be performed using the following grading scale:
  N0 - No nerve damage N1 - Minor: sensory paresthesia N2 - Major: complete sensory anesthesia N3 - Complete: complete motor deficit with or without paresthesia N4 - CRPS: Complex Regional Pain Syndrome
glucose | 12 hours after surgery
  blood glucose level
glucose | 24 hours after surgery
  blood glucose level
glucose | 48 hours after surgery
  blood glucose level

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes